CLINICAL TRIAL: NCT04635475
Title: Return to Learn Implementation Bundle for Schools (RISE) After Youth Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Monica Vavilala, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008181; 1R49CE003087-01 (NIH)
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Testing RISE bundle to improve RTL care after concussion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Consented parents of a concussed high school student who will receive CDC Head's UP Concussion Guidelines during a five week program. 75 Participants.
- Intervention Group (Experimental): Consented parents of a concussed high school student who will receive the CDC Head's Up Concussion Guidelines and intervention RTL Student Protocol during a five week program. 75 Participants.
  Interventions: Behavioral: RISE Bundle

INTERVENTIONS:
Behavioral: RISE Bundle — Toolkit to build capacity where students receive education and provide symptom based and tailored accommodations after concussion
  Arms: Intervention Group

SUMMARY:
Using the Consolidated Framework for Implementation Research, as our overarching conceptual framework, this translational 2 ½ year pragmatic RCT uses a clustered, stepped wedge design to test the effectiveness of a school-based (unit of analysis) implementation strategy (project intervention) called RISE (Return to Learn Implementation bundle for schools) on evidence-based practice (RTL protocol implementation; main outcome) and student outcomes (i.e., days to RTL start after diagnosis) after youth concussion. The central hypothesis is that schools in the intervention condition receiving the RISE implementation bundle (toolkit plus school support) will have more complete and sustainable RTL protocols, and better student outcomes compared to schools in control condition who receive only written RTL protocol information. As rural and low SES schools are particularly likely to struggle to implement RTL protocols,19,25 we specifically examine RISE implementation and barriers to implementation related to school demographic characteristics related to health equity. The school characteristics we examine are rurality, primary language, racial and ethnic mix, and free/reduced-cost lunch.

DETAILED DESCRIPTION:
As you are aware, COVID caused us to consider how to complete this project and answer the scientific questions posed in the Specific Aims. The investigators considered shifting the RTL project to a later time and switching with another project but this would not have worked for the other project.

To solve this challenge of impact of school changes, the investigators convened with the project advisory board for consultation, consulted the research core at HIPRC and contacted the participants who were to have been participants in the randomized controlled trial. 19 of the 24 schools responded. From this work, the investigators agreed that since the school context has changed to either home online or hybrid mode, that students with concussion who are the recipients of the intervention should not be deprived of an intervention that is potentially beneficial.

The investigators have therefore made the following adaptations that retained the specific aims and central hypothesis that school context capacity can be strengthened to provide tailored student-centered RTL care and improve outcomes for students with a concussion.

To this end, the investigators are considering "school" wherever students are receiving an education. The investigators will recruit subjects who are currently largely coordinating education due to COVID, work with their schools, and recruit nationally. These adaptations will require a sample size of a total of 150 high school students with recent concussion (75 intervention [Group A: RISE bundle + CDC information], 75 controls [Group B: CDC information only]) who will be recruited using social media and other platforms.

There are some advantages to this design: 1) The investigator's intervention materials will now be able to be translated to Spanish due to adaptations, 2) This project will reach more particpants in rural and from disadvantaged backgrounds, 3) Communications between particpants and schools will be enhanced.

Given return to school, we have reverted to the stepped wedge study design in WA state.

ELIGIBILITY:
Inclusion Criteria: Public high school student, grade 9th - 12th who has sustained a concussion.

* High School Student between the age of 14-19, who attends in person, online, or a hybrid academic platform, and the concussion did not include an acute care hospital course greater than 48 hours.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
RTL OUTCOMES - Symptom | 5 week
  Tracking children's symptoms over a five-week period of time. Parental completion of 4 - week symptom checklist 100% completion of weekly symptom checklist resulting in 20% fewer symptoms for the intervention group.

SECONDARY OUTCOMES:
RTL OUTCOMES - Academic Success | 5 week
  Outcome measures to assess academic success. Parental completion of CLASS survey weeks 2 and 4 resulting in a 20 % less decline Intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Monica S Vavilala, MD, Principal Investigator — University of Washington
Locations (1):
- HIPRC, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data

REFERENCES:
- See also: Consolidated Framework — https://implementationscience.biomedcentral.com/articles/10.1186/1748-5908-4-50